CLINICAL TRIAL: NCT04797039
Title: MRI-Guided Cryoablation for Focal Native Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Woodrum, M.D, Ph.D, Principal Investigator, Mayo Clinic
Other Study IDs: 20-003822
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Primary Malignant Neoplasm of Prostate (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Cryosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MR guided cryoablation: Focal MR guided cryoablation for low- to intermediate-grade prostate cancer
  Interventions: Procedure: MR guided cryoablation

INTERVENTIONS:
Procedure: MR guided cryoablation — MR guided cryoablation of focal biopsy proven prostate cancer
  Other Names: cryoablation

SUMMARY:
The purpose of this research is to collect data about the MRI cryoablation procedure your doctor(s) would normally perform in order to treat the participants focal prostate cancer and to evaluate the participants condition after the participants treatment is performed.

Participants have been asked to take part in this research because the participants have been diagnosed with prostate cancer and scheduled to have an ablation procedure.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate MR-guided cryoablation of biopsy proven prostate tumors using the Galil MRI-compatible cryoablation system. The system has been approved by the United States Food and Drug Administration (FDA) for soft tissue ablation and has been utilized successfully at Mayo. All procedures will be performed according to approved indications. the investigators wish to monitor the technique and collect data at the participants follow-up visits.

The study only collects data about the MRI-guided cryoablation procedure the participants doctor(s) would normally perform in order to treat the participants focal prostate cancer and to evaluate the participants condition after there treatment is performed. The participants doctor will advise the participants when the participants should return for follow-up visits. These visits will be according to the participants doctor's standard of care; usually return visits are at 3-6months, 12 months, 24 months, 36 months, 48 months and 60 months after the procedure, although the participants doctor may ask that the participants return for more frequent visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with "biopsy proven" Gleason7 prostate cancer referred to Urology and/or Interventional Radiology for treatment
* Surgery and/or Radiation is not a desirable alternative therapy at the time of enrollment
* Tumor size is < 2 cm at its largest diameter
* Tumor does not encompass the rectal wall or external urethral sphincter
* Patient is able to undergo MRI

Exclusion Criteria:

•

Ages: 30 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male population 50-100 years old with biopsy confirmed localized low- to intermediate-grade cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Technical success of the MR-guided cryoablation | Will assess for 5 years with interval assessment each year
  Determine the technical success of the MR-guided cryoablation as measured by complete target lesion ablation.
Safety of the MR-guided cryoablation | Will assess for 5 years with interval assessment each year
  Determine safety of the MR-guided cryoablation using continuous MR imaging during the procedure.
Examine short term tumor recurrence | Will assess for 5 years with interval assessment each year
  Examine short term tumor recurrence over 6 months with contrast enhanced MRI and as required MR or U/S guided biopsy of prostate bed if PSA biochemical recurrence.

SECONDARY OUTCOMES:
MR procedure time. | Will assess for 5 years with interval assessment each year
  We will examine the time for each step in the process to create a stream-lined process and minimize MR procedure time.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials